CLINICAL TRIAL: NCT02214693
Title: A Clinical Study to Investigate the Pharmacokinetics/Pharmacodynamics and Tolerability of DA-1229(Evogliptin) Tablet in Renal Impaired Patients
Brief Title: PK//PD/Tolerability Study of DA-1229(Evogliptin) in Renal Impaired Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: DA1229_RI_I
Record Dates: First submitted 2014-08-11; First posted 2014-08-12 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Renal Impairment
Keywords: patients
MeSH Terms: conditions — Renal Insufficiency | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1(Severe decrease in GFR) (Experimental): Severe decrease in GFR
  Interventions: Drug: DA-1229
- Group 2(Moderate decrease in GFR) (Experimental): Moderate decrease in GFR
  Interventions: Drug: DA-1229
- Group 3(Mild decrease in GFR) (Experimental): Mild decrease in GFR
  Interventions: Drug: DA-1229
- Group 4(Normal GFR) (Experimental): Normal GFR
  Interventions: Drug: DA-1229

INTERVENTIONS:
Drug: DA-1229
  Other Names: Evogliptin

SUMMARY:
This is a clinical study to investigate the pharmacokinetics/pharmacodynamics and tolerability of DA-1229(Evogliptin) tabletin renal impaired patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 70
* Weights between 50 and 90kg(Female : 40 and 90kg)
* Volunteer who totally understands the progress of this clinical trials, makes decision by his free will, and signed a consent form to follow the progress
* Stable results of estimated GFR in 4 months recently

Exclusion Criteria:

* Volunteer who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, Neurology, immunology, pulmonary, endocrine, hematooncology, cardiology, mental disorder)
* Volunteer who had drug(DPP-4 inhibitor) hypersensitivity reaction
* Volunteer who already participated in other trials in 2 months
* Volunteer who had whole blood donation in 2 months, or component blood donation in 1 months or transfusion

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Area Under Curve(AUC) last | Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72, 96, 120h post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Seoul National University Hospital, Seoul, South Korea